CLINICAL TRIAL: NCT02929797
Title: A Randomized, Double Blinding, Placebo-Controlled Clinical Trials of CD8+NKG2D+ AKT Cell Immunotherapy to the Pancreatic Cancer Patients Treated With Adjuvant Chemotherapy
Brief Title: Immunotherapy of CD8+NKG2D+ AKT Cell With Chemotherapy to Pancreatic Cancer
Acronym: AKT
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Shanghai iCELL Biotechnology Co., Ltd, Shanghai, China (Industry)
Responsible Party: Principal Investigator, Hongxia Wang, Deputy Director of Oncology, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CD8+NKG2D+ AKT
Record Dates: First submitted 2016-10-07; First posted 2016-10-11 (Estimated); Last update posted 2016-10-11 (Estimated); Status verified 2016-10

CONDITIONS: Pancreatic Ductal Adenocarcinoma
Keywords: pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AKT + gemcitabine (Experimental): gemcitabine dose 1000mg/M^2, d1,8,15，q4w ×6 AKT 5*10^8/M^2, d16,q4w ×6 Drug: gemcitabine Biological: AKT, CD8+NKG2D+ AKT Cell
  Interventions: Biological: CD8+NKG2D+ AKT Cell; Drug: Gemcitabine
- gemcitabine (Active Comparator): gemcitabine hydrochloride dose 1000mg/M2 d1,8,15，q4w ×6 Drug: gemcitabine
  Interventions: Drug: Gemcitabine

INTERVENTIONS:
Biological: CD8+NKG2D+ AKT Cell — AKT: CD8+NKG2D+ AKT cell
  Other Names: AKT
  Arms: AKT + gemcitabine
Drug: Gemcitabine — gemcitabine
  Other Names: GEM

SUMMARY:
A Prospective Study on the Efficacy and Safety of CD8+NKG2D+ AKT cell immunotherapy to the pancreatic cancer patients treated with adjuvant chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* 1. Diagnosed as stage II-III pancreatic ductal adenocarcinoma patients by pathologic histology;
* 2. Pancreatic cancer after radical resection;
* 3. Eastern Cooperative Oncology Group Performance Status less than 2;
* 4. Without radiotherapy or neoadjuvant chemotherapy;
* 5. The man or the gestation and lactation women Age between 18 to 80 years old;
* 6. Bone marrow functioned well: ANC more than 1.5*10^9/ L, PLT more than 100*10^9/LHgb more than 9 g/dL;
* 7. Blood biochemical indicators: AST（SGOT）less than 1.5 ULNALT（SGPT）less than 1.5 ULN, TBIL less than 1.5 ULN;
* 8. PT and PPT are in normal ranges;
* 9. Three months prior to clinical research did not receive any other clinical research trials;
* 10. patients are voluntary, and willing to sign informed consent.

Exclusion Criteria:

* 1. Patients with other malignant tumors in the past five years;
* 2. Active viral or bacterial infection and cannot be controlled with appropriate anti-infection treatment;
* 3. Known as HIV infection, active hepatitis B virus or hepatitis C virus infection;
* 4. Known allergy to any kind of component of study drugs;
* 5. History of connective tissue disease(Such as lupus, scleroderma, nodular arteritis);
* 6. Patients with a history of interstitial pneumoniaSlowly progressive difficulty in breathing and hoose Sarcoidosissilicosis Fibrose pulmonaire idiopathiquehylactic pneumonia or A variety of allergy;
* 7. Suffering from mental illness or other illness, such as heart or lung disease, diabetes, etc. that can not be controlled, and can not cope with study treatment and monitoring requirements;
* 8. At the same time Patients participate in any other use of interventional medicine clinical research or checkers.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-08 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | 1 year

SECONDARY OUTCOMES:
Overall Survival | 3 years
immune indices | 1 year
Quality of life | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: hongxia Wang, Dr., Principal Investigator — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Locations (2):
- China (2):
  - Shanghai General Hospital, Shanghai, Shanghai Municipality
  - Shanghai General Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: Undecided